CLINICAL TRIAL: NCT05985278
Title: Clinical Application of Lutetium [177Lu]-Catalase in Tumor Radionuclide Therapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021KT90
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Advanced Malignant Neoplasm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [ Lu-177]-Catalase (Experimental): Participants received [ Lu-177]-Catalase intratumoral injection
  Interventions: Drug: [ Lu-177]-Catalase

INTERVENTIONS:
Drug: [ Lu-177]-Catalase — [ 177Lu]-Catalase is administered by intratumoral puncture every four weeks, and the specific dose is related to the size of the tumor

SUMMARY:
The purpose of this study is to evaluate the retention in tumour and distribution behavior of [Lu-177]-Catalase after intratumoral injection,and preliminary evaluation the efficacy and safety of [Lu-177]-Catalase.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 2-week screening period to determine eligibility for study entry. At day1, patients who meet the eligibility requirements will be intratumoral injection the [Lu-177]-Catalase.The efficacy evaluation will be conducted at one month p.i., whether to continue intratumoral injection the [Lu-177]-Catalase, depending on the patient's efficacy and safety results.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 18-70 years; ECOG score 0 or 1;
2. Patients with advanced malignant tumors, such as liver cancer, ovarian cancer, prostate cancer, and so on, clearly diagnosed by pathology and/or cytology;
3. Patients with advanced solid tumors who have failed or cannot tolerate standard treatment;
4. Expected survival of more than 3 months;
5. According to the solid tumor efficacy evaluation criteria , the patient had at least one measurable or evaluable tumor lesion with the longest diameter ≥10 mm at baseline (in the case of lymph nodes, the short diameter ≥15 mm). This lesion is suitable for intratumoral injection (the length of the lesion is at least 1 cm or equal).
6. Blood routine and liver and kidney function meet the following criteria: Blood routine: WBC≥4.0×109L or neutrophil ≥1.5×109L, PLT≥100×109/L, Hb≥90g/L; PT or APTT≤1.5ULN; Liver and kidney function: T-Bil≤1.5×ULT(upper limit of normal),ALT/AST≤2.5ULN or ≤5×ULT(subjects with liver metastasis), ALP≤2.5ULN(ALP≤ 4.5ULN if there is bone metastasis or liver metastasis); BUN≤1.5×ULT, SCr≤1.5×ULT;
7. Women must use effective contraception during the study period and for 6 months after the study (effective contraception means sterilization, intrauterine hormone devices, condoms, contraceptives/pills, abstinence or partner vasectomy, etc.); Men should consent to subjects who must use contraception during the study period and for 6 months after the end of the study period;
8. Can understand and voluntarily sign informed consent, compliance is good

The Exclusion Criteria:

1. Severe abnormal liver and kidney function;
2. Pregnant, pregnant and lactating women;
3. Can not lie flat for half an hour;
4. Refuse to join the clinical investigator;
5. Suffering from claustrophobia or other mental illness;
6. Other conditions deemed unsuitable for participation in the trial by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The absorbed radiation dose of tumor and normal organs | From first dose of study drug through 8 weeks post dose
  Calculation of effective absorbed dose of tumor in situ injection

SECONDARY OUTCOMES:
Preliminary efficacy of [ Lu-177]-Catalase based on tumor response | From first dose of study drug through 8 weeks post dose
  Tumor volume based on RECIST 1.1.

OTHER OUTCOMES:
Adverse events for [ Lu-177]-Catalase | From first dose of [ Lu-177]-Catalase through 8 weeks post dose.
  Occurrence of adverse events for [ Lu-177]-Catalase

CONTACTS AND LOCATIONS:
Locations (1):
- Zhi Yang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided